CLINICAL TRIAL: NCT06203431
Title: A Multicenter, Randomized, Double-blind, Etomidate-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of ET-26 for Induction of General Anesthesia in Subjects Undergoing Elective Surgery
Brief Title: A Trial to Evaluate the Efficacy and Safety of Methoxyetomidate Hydrochloride for Injection (ET-26) for the Induction of General Anesthesia in Elective Surgery Subjects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-26-HCl-301
Record Dates: First submitted 2023-12-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia Induction
Keywords: Elective Surgery, Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug ET-26 (Experimental)
  Interventions: Drug: ET-26
- Drug Etomidate (Active Comparator)
  Interventions: Drug: Etomidate Injectable Emulsion

INTERVENTIONS:
Drug: ET-26 — freeze-dried powder injection，The initial dose is 0.8 mg/kg, with an additional 50% starting dose if needed. single dose, Infusion time was 60s ± 5s.
  Arms: Drug ET-26
Drug: Etomidate Injectable Emulsion — lipid emulsion ，The initial dose is 0.3 mg/kg, with an additional 50% starting dose if needed.single dose, Infusion time was 60s ± 5s.
  Arms: Drug Etomidate

SUMMARY:
This is a multicenter, randomized, double-blind, etomidate-controlled phase III clinical trial. The primary objective is to compare the efficacy and safety between ET-26 and etomidate in the induction of general anesthesia in subjects undergoing elective surgery, so as to provide a reference for the marketing registration of methoetomidate hydrochloride for injection.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients requiring tracheal intubation under general anesthesia for Non-emergency, non-cardiothoracic, non-extracranial elective surgery estimated operation duration ≥ 0.5h;
2. Age ≥ 18 and ≤ 70 years old, gender is not limited;
3. ASA（American Society of Anesthesiologists） Class I-II;
4. Body mass index (BMI) 18 ~ 30 kg/m2 (including boundary value);
5. Serum cortisol concentration test is normal or abnormal but judged no clinical significance by the investigator;
6. Vital signs during screening: respiratory rate≥ 10 and ≤ 24 breaths /minute; When breathing air, pulse oxygen saturation (SpO2)≥95%; Systolic blood pressure (SBP) ≥ 90mmHg and ≤160mmHg; diastolic blood pressure (DBP) ≥ 60mmHg and ≤100mmHg; heart rate (ECG results) ≥ 55 and ≤ 100 beats/min;
7. Subjects must understand the procedures and methods of this study and be willing to sign informed consent and strictly abide by this trial protocol to complete the study.

Exclusion Criteria:

1. Subjects with contraindications to general anesthesia or previous history of anesthesia accidents, and other systemic medical history that increases the risk of anesthesia;
2. Known or suspected family history of malignant hyperthermia;
3. Known or suspected of being allergic or contraindicated to the procedural medication prescribed in each component or regimen of the experimental drug, suspected of epilepsy or severe liver and kidney dysfunction;
4. Difficulty in intubation or ventilation is expected (Modified Mallampati Score of Ⅲ and Ⅳ);
5. Presence of any of the following respiratory management risks before/at screening: 1) history of asthma, stridor; 2) Patients with sleep apnea syndrome;
6. Any of the following drugs or treatments were used prior to screening: 1) those who participated in any drug clinical trial within 1 month prior to screening; 2) Have used drugs or treatments that affect cortical function within 3 days before screening; 3) Use of drugs that may affect the QT interval within 2 weeks prior to screening;
7. The laboratory examination indicators during the screening period meet the following standards:

1) AST and /or ALT ≥ 3×ULN; 2)TBIL≥1.5×ULN； 3) Hb≤90 g/L (and no blood transfusion within 14 days); 4)ANC≤1.5×109/L； 5)PLT≤80×109/L； 6) Blood Serum creatinine ≥1.5×ULN; 8. Pregnant and lactating women; the reluctance of fertile women or men to use contraception throughout the trial; subjects (including male subjects) who had pregnancy plans within three months of the trial; 9. Subjects who have any other factors deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of anesthesia induction | within 7minutes after injection
  modified observer's assessment of alert≤1 (only one additional dose was allowed) and endotracheal intubation was completed within 7 minutes from the beginning of study drug infusion, and no remedial drugs were used

SECONDARY OUTCOMES:
Time to loss of consciousness | Time from first administration of study drug to MOAA/S（modified observer's assessment of alert）≤1,every 1 minute ±5 seconds, within 3 minutes after injection
The percentage of time between 40≤BIS（Bispectral index）≤60 | During the period from the initial administration to the successful intubation of the tracheal tube,every 1 minute±20 seconds, within 7minutes after injection
The percentage of subjects with eyelash reflexes disappearing | within 3 minutes after injection
time required to achieve eyelash reflex disappearance | within 3 minutes after injection
the use of investigational drugs and remedial drugs | Induction period of anesthesia,within 7minutes after injection
Proportion of subjects using remedial sedatives | Induction period of anesthesia,within 7minutes after injection
The time to successfully intubate | within 7minutes after injection
intubation reaction | within 5 minutes after successful intubation
  Whether coughing, body movement reaction
Changes of BIS（Bispectral index） within 30 minutes after endotracheal intubation successfully (such as the time percentage between BIS 40 and BIS 60) | 30 minutes after successful intubation
Anesthesiologists' satisfaction scores on the transition between induction and maintenance of anesthesia. | immediately after surgery
  The anesthesiologist's satisfaction score for the connection between induction of anesthesia and maintenance of anesthesia, on a scale of 10, 0 being very dissatisfied and 10 being very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: JIN LIU, Medicine Doctor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China